CLINICAL TRIAL: NCT00317304
Title: Mindfulness Based Stress Reduction for Hot Flashes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, James Carmody, Study Principle Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT002910-01 (NIH); R21AT002910-01 (NIH)
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Hot Flashes; Stress
Keywords: Hot flashes; vasomotor symptoms; menopause; mindfulness based stress reduction; meditation
MeSH Terms: conditions — Hot Flashes | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MBSR (Experimental)
  Interventions: Behavioral: Mindfulness-based stress reduction

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction — MBSR is an 8-week group-based program of training in mindfulness and its application to the stresses and challenges of everyday life
  Other Names: MBSR

SUMMARY:
Stress appears to be related to hot flash frequency and intensity, and the degree of distress that women experience from their hot flashes appears to be related to their coping resources. This trial is a pilot study to test the effect of participation in a mindfulness-based stress reduction program on hot flash frequency and intensity, as well as menopause-related quality of life.

DETAILED DESCRIPTION:
The majority of women experience vasomotor symptoms (VMS) such as hot flashes (HF) and night sweats as they transition through menopause, and a substantial minority experience considerable distress and diminished role functioning. Until recently most women found relief through hormone therapy (HT), but concern about the health risks associated with HT has left women with few effective and safe choices for relief from their symptoms other than their own coping strategies. A variety of results from both population and laboratory studies suggest that stress and HF are correlated and that HF are more severe in women with lower coping abilities, but evidence is far from conclusive. Consequently, investigators have called for trials to evaluate the effect of stress reduction interventions on HF. Mindfulness-Based Stress Reduction (MBSR) is a widely available manualized program shown to be an effective adjunctive intervention in reducing medical symptoms and psychological distress for a wide range of stress-related disorders. In a small preliminary study using MBSR we found reductions in HF severity scores and increases in menopause-related quality of life (QOL). This R21 proposal is for a pilot randomized trial of MBSR compared to a wait-list control group for 120 menopausal women experiencing seven or more HF/day of moderate to severe intensity. It aims to:

1. assess feasibility of recruitment, adherence to program intervention, and compliance with assessment instruments in preparation for a larger RCT; and
2. provide preliminary estimates of efficacy of the effects of MBSR in reducing self-reported HF frequency and intensity and improving QOL.

In addition, we will use sternal skin conductance as an established objective measure of VMS in a subgroup of 15 women in each arm to test feasibility and obtain information on how objectively measured HF are related to self-reported HF in this setting. Women will be assessed at baseline, at the end of the eight-week MBSR course, and at three months after the end of the course. A secondary aim is to explore whether treatment group differences of HF frequency and intensity and QOL are explained by changes in perceived stress, health-related locus of control and mindfulness. It is anticipated that results from this pilot study will provide data needed to plan a larger more definitive randomized trial on the effect of MBSR on HF frequency and intensity and on the ability to cope with these symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Average of 5+ hot flashes per day
* No menses in prior 3 months
* Ages between 40 and 69 years
* English speaking
* Access to a telephone
* Availability for the entire study period
* Agree to maintain usual diet
* Agree to maintain usual exercise habits
* Consent to the study

Exclusion Criteria:

* Psychiatric illness
* Illness with less than one year life expectancy
* Alcohol use ≥ 2 drinks per day
* Current substance abuse or addiction
* Use of selective estrogen receptor modulator (SERM) medications within the past 3 months
* Use of HT within the past 3 months
* Currently pregnant or breastfeeding
* Ongoing mindfulness meditation practice

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2005-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Hot flash frequency and intensity | Baseline, 8 weeks, 24 weeks

SECONDARY OUTCOMES:
Menopause-related quality of life | Baseline, 8 weeks, 24 weeks
Hot Flash-Related Daily Interference Scale | Baseline, 8 weeks, 24 weeks
Women's Health Initiative (WHI) Insomnia Rating Scale | Baseline, 8 weeks, 24 weeks
5 factor of Mindfulness questionnaire | Baseline, 8 weeks, 24 weeks
Health locus of control | Baseline, 8 weeks, 24 weeks
Perceived stress | Baseline, 8 weeks, 24 weeks
Dietary intake | Baseline, 8 weeks, 24 weeks
Compliance with intervention conditions | Baseline, 8 weeks, 24 weeks
HADS | Baseline, 8 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James Carmody, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Carmody JF, Crawford S, Salmoirago-Blotcher E, Leung K, Churchill L, Olendzki N. Mindfulness training for coping with hot flashes: results of a randomized trial. Menopause. 2011 Jun;18(6):611-20. doi: 10.1097/gme.0b013e318204a05c. PMID 21372745